CLINICAL TRIAL: NCT02175680
Title: A Phase 2b Study to Assess Suppression of HIV-1 Replication Following Substitution of Stable Combination Antiretroviral Therapy With a PRO 140 (Monoclonal CCR5 Antibody) Monotherapy in Adult Subjects With HIV-1 Infection
Brief Title: Treatment Substitution With PRO 140 Monotherapy in Adult Subjects With HIV-1 Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CytoDyn, Inc. (Industry)
Collaborators: Amarex Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO 140_CD 01
Record Dates: First submitted 2014-06-24; First posted 2014-06-26 (Estimated); Results first posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-03

CONDITIONS: HIV; Human Immunodeficiency Virus
Keywords: HIV-1; HIV; Treatment Substitution; PRO 140; PRO140; CytoDyn; Amarex
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — leronlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PRO 140 (Experimental): PRO 140 350mg weekly SQ injection.
  Interventions: Drug: PRO 140; Other: Historical data

INTERVENTIONS:
Drug: PRO 140 — CCR5 Antagonist
  Other Names: PRO 140 350mg
Other: Historical data — Historical data (i.e., time to HIV-1 RNA viral load > 500 copies/mL of 29 days).

SUMMARY:
This study is a Phase 2b study designed to evaluate the efficacy, safety, and tolerability of PRO 140 monotherapy for the maintenance of viral suppression in subjects who are stable on combination antiretroviral therapy.

Consenting subjects will be shifted from their combination antiretroviral regimen to PRO 140 monotherapy for 12 weeks. Total treatment duration with PRO 140 will be 14 weeks with the one week overlap of existing retroviral regimen and PRO 140 at the beginning of the study treatment, and one week overlap at the end of the treatment in subjects who do not experience virologic failure.

DETAILED DESCRIPTION:
This study is a Phase 2b, multi-center study designed to evaluate the efficacy, safety, and tolerability of PRO 140 monotherapy for the maintenance of viral suppression in patients who are stable on combination antiretroviral therapy.

Patient enrollment will be staggered in this study to facilitate adequate safety monitoring. A lead cohort will include 12 subjects. Enrollment of additional 28 subjects will not be initiated until it is approved by the independent Data Monitoring Committee (DMC).

Consenting patients will be shifted from combination antiretroviral regimen to PRO 140 monotherapy for 12 weeks. Total treatment duration with PRO 140 will be up to 14 weeks with the one week overlap of existing retroviral regimen and PRO 140 at the beginning of the study treatment and also one week overlap at the end of the treatment in subjects who do not experience Virologic Failure.

PRO 140 will be administered as a 350 mg subcutaneous injection weekly for up to 14 weeks. Study participants will be monitored for viral rebound on a weekly basis following initiation of PRO 140 monotherapy and will re-initiate their previous antiretroviral regimen if plasma HIV-1 RNA levels rise above 400 copies/ml on two consecutive blood draws at least 3 days apart.

The study will have three phases: Screening Phase, Treatment Phase and Follow-up Phase.

The primary objective is to assess efficacy of PRO 140 monotherapy for the maintenance of viral suppression following substitution of antiretroviral therapy in patients who are stable on combination antiretroviral therapy.

The secondary objective of the trial is to assess the clinical safety and tolerability parameters following substitution of antiretroviral therapy in patients who are stable on combination antiretroviral therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, age ≥18 years
2. Exclusive CCR5-tropic virus at Screening Visit as determined by Trofile™ DNA Assay
3. On stable antiretroviral therapy for last 12 months
4. Subject has two or more potential alternative antiretroviral regimen options to consider.
5. No documented detectable viral loads (HIV-1 RNA <50 copies/ml) within the last 12 months prior to Screening Visit
6. Nadir CD4 cell count of >200 cells/mm3

Exclusion Criteria:

1. CXCR4-tropic virus or dual/mixed tropic (R5X4) virus determined by the Trofile™ DNA Assay at the Screening Visit
2. Hepatitis B infection as manifest by the presence of Hepatitis B surface antigen (HBsAg)
3. Any acquired immune deficiency syndrome (AIDS)-defining illness according to the 1993 Centers for Disease Control and Prevention (CDC) AIDS surveillance definition
4. Prior use of any entry, attachment, CCR5 co-receptor, or fusion inhibitor, including PRO 140.
5. Any other clinical condition that, in the Investigator's judgment, would potentially compromise study compliance or the ability to evaluate safety/efficacy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2014-04-16 (Actual); Primary Completion 2015-02-02 (Actual); Study Completion 2015-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Lalezari, MD, Principal Investigator
Locations (1):
- Quest Clinical Research, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chang XL, Reed JS, Webb GM, Wu HL, Le J, Bateman KB, Greene JM, Pessoa C, Waytashek C, Weber WC, Hwang J, Fischer M, Moats C, Shiel O, Bochart RM, Crank H, Siess D, Giobbi T, Torgerson J, Agnor R, Gao L, Dhody K, Lalezari JP, Bandar IS, Carnate AM, Pang AS, Corley MJ, Kelly S, Pourhassan N, Smedley J, Bimber BN, Hansen SG, Ndhlovu LC, Sacha JB. Suppression of human and simian immunodeficiency virus replication with the CCR5-specific antibody Leronlimab in two species. PLoS Pathog. 2022 Mar 31;18(3):e1010396. doi: 10.1371/journal.ppat.1010396. eCollection 2022 Mar. PMID 35358290

RESULTS

PARTICIPANT FLOW:
Groups:
- PRO 140 350 mg Weekly SQ Injection: Subject enrollment was staggered in this study to facilitate adequate safety monitoring. The lead cohort included 12 subjects. Enrollment of an additional 28 subjects was initiated after approval by the independent Data Monitoring Committee (iDMC).Consenting subjects were shifted from combination antiretroviral regimen to PRO 140 monotherapy for 12 weeks. Total treatment duration with PRO 140 was up to 14 weeks, with one (1) week overlap of existing retroviral regimen and PRO 140 at the beginning end of the treatment in subjects who did not experience Virologic Failure. PRO 140 was administered as a 350 mg subcutaneous injection weekly for up to 14 weeks. Study participants were monitored for viral rebound on a weekly basis following initiation of PRO 140 monotherapy and re-initiated their previous antiretroviral regimen if plasma HIV-1 RNA levels were ≥ 400 copies/ml on two (2) consecutive blood draws at least three (3) days apart.
Period: Overall Study
Arm/Group | PRO 140 350 mg Weekly SQ Injection
Started | 43
Completed | 41
Not Completed | 2
Not completed — non-compliance | 1
Not completed — other non-medical reason | 1

BASELINE CHARACTERISTICS:
Groups:
- PRO 140: PRO 140 350mg weekly SQ injection.
  PRO 140 350mg weekly SQ injection.: CCR5 Antagonist
Arm/Group | PRO 140
Number analyzed (Participants) | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.1 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 34
  More than one race | 0
  Unknown or Not Reported | 5
Time since HIV Diagnosis (Years) [Mean (Standard Deviation); unit: years] | 18.8 (9.5)

OUTCOME MEASURES:

1. Primary Outcome: Time to Virologic Failure After Initiating PRO 140 Monotherapy.
Description: Time to virologic failure after initiating PRO 140 monotherapy. Virologic failure was defined as two (2) consecutive HIV-1 RNA levels of ≥ 400 copies/mL.
Time Frame: From initiation of PRO 140 monotherapy through week 14 or virological failure
Population: Per Protocol population
Measure: Mean (Standard Deviation); unit: days
Groups:
- PRO 140 350 mg: PRO 140 350 mg weekly SQ injection.
Arm/Group | PRO 140 350 mg
Number analyzed (Participants) | 41
days | 70.71 (23.14)
Statistical Analysis 1: Comparison: PRO 140 350 mg; Test type: Superiority; p < 0.0001, Wilcoxon Rank Sum; The time to Virologic Failure for the subjects treated with PRO 140 monotherapy was compared to historical data; The median time to Virologic Failure for historical controls was 29 days

2. Secondary Outcome: Proportion of Subjects With Virologic Failure
Description: Proportion of Participants with Virologic Failure after initiating PRO 140 monotherapy at or prior to Week 14.
Time Frame: From initiation of PRO 140 monotherapy through week 14
Population: Per Protocol
Measure: Number; unit: poportion of subjects
Arm/Group | PRO 140 350 mg
Number analyzed (Participants) | 41
poportion of subjects | 0.439

3. Secondary Outcome: Mean Change From Baseline in Viral Load
Description: Mean change in Viral Load (HIV-1 RNA levels - log 10 copies/ml)), at each visit within the 14-week treatment phase.
Time Frame: From initiation of PRO 140 monotherapy through week 14
Population: Per Protocol population
Measure: Mean (Standard Deviation); unit: log 10 copies/mL
Groups:
- PRO 140: PRO 140 350mg
Arm/Group | PRO 140
Number analyzed (Participants) | 41
log 10 copies/mL
  T2 (Week 2): number analyzed (Participants) | 40
  T2 (Week 2) | 0.10 (0.71)
  T3 (Week 3) | 0.01 (0.74)
  T4 (Week 4) | -0.13 (0.74)
  T5 (Week 5): number analyzed (Participants) | 40
  T5 (Week 5) | -0.25 (1.04)
  T6 (Week 6) | -0.76 (1.39)
  T7 (Week 7): number analyzed (Participants) | 39
  T7 (Week 7) | -0.88 (1.53)
  T8 (Week 8): number analyzed (Participants) | 35
  T8 (Week 8) | -0.72 (1.37)
  T9 (Week 9): number analyzed (Participants) | 33
  T9 (Week 9) | -0.84 (1.37)
  T10 (Week 10): number analyzed (Participants) | 28
  T10 (Week 10) | -0.71 (1.36)
  T11 (Week 11): number analyzed (Participants) | 28
  T11 (Week 11) | -0.81 (1.37)
  T12 (Week 12): number analyzed (Participants) | 27
  T12 (Week 12) | -0.91 (1.50)
  T13 (Week 13): number analyzed (Participants) | 23
  T13 (Week 13) | -0.44 (1.12)
  T14 (Week 14): number analyzed (Participants) | 8
  T14 (Week 14) | -0.37 (1.09)

4. Secondary Outcome: Change in Viral Load at the Last Virologic Failure Visit.
Description: Mean Change from Baseline in viral load at the last virologic failure visit from Week 1 to Week 14. VF can occur at any time during the treatment phase from week 1 to week 14. Subjects who experience Virologic Failure will be followed up every 4 weeks until the viral load suppression is achieved (i.e., plasma HIV-1 RNA levels to return back to <50 copies/mL)
Time Frame: From baseline to virologic failure visit (VF). VF can occur at any time from Week 1 to Week 14.
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: log 10 copies/ml
Arm/Group | PRO 140 350 mg Weekly SQ Injection
Number analyzed (Participants) | 40
log 10 copies/ml | -1.78 (1.93)

5. Secondary Outcome: Mean Change in CD4 Cell Count by Visit
Description: Mean change in CD4 cell count, at each visit within the 14-week treatment phase
Time Frame: From baseline (week 2) through week 14
Population: Per protocol
Measure: Mean (Standard Deviation); unit: cells/mm^3
Groups:
- PRO 140: PRO 140 350mg/mL
Arm/Group | PRO 140
Number analyzed (Participants) | 41
cells/mm^3
  T2 (Week 2): number analyzed (Participants) | 40
  T2 (Week 2) | 32.05 (132.92)
  T3 (Week 3): number analyzed (Participants) | 14
  T3 (Week 3) | -33.14 (137.05)
  T4 (Week 4): number analyzed (Participants) | 40
  T4 (Week 4) | -12.78 (137.37)
  T5 (Week 5): number analyzed (Participants) | 12
  T5 (Week 5) | 33.42 (130.88)
  T6 (Week 6): number analyzed (Participants) | 38
  T6 (Week 6) | -3.26 (125.78)
  T7 (Week 7): number analyzed (Participants) | 10
  T7 (Week 7) | 47.50 (190.10)
  T8 (Week 8): number analyzed (Participants) | 34
  T8 (Week 8) | -55.09 (157.21)
  T9 (Week 9): number analyzed (Participants) | 8
  T9 (Week 9) | 47.25 (95.64)
  T10 (Week 10): number analyzed (Participants) | 28
  T10 (Week 10) | -6.82 (140.34)
  T11 (Week 11): number analyzed (Participants) | 6
  T11 (Week 11) | -29.83 (218.64)
  T12 (Week 12): number analyzed (Participants) | 25
  T12 (Week 12) | 16.52 (143.91)
  T13 (Week 13): number analyzed (Participants) | 16
  T13 (Week 13) | -0.44 (95.54)
  T14 (Week 14): number analyzed (Participants) | 7
  T14 (Week 14) | -59.03 (56.50)
  VF (Viral failure): number analyzed (Participants) | 17
  VF (Viral failure) | 18.41 (113.99)

6. Secondary Outcome: Mean Change in CD4 Cell Count
Description: Change from baseline in CD4 cell count, within the 14-week treatment phase
Time Frame: From baseline (week 2) to last visit
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: cells/mm^3
Groups:
- PRO 140: PRO140 350 mg
Arm/Group | PRO 140
Number analyzed (Participants) | 41
cells/mm^3 | 18.97 (114.08)

7. Secondary Outcome: Q1 QOL Health Status
Description: Quality of Life Q1 Current General Health Status, is collected from base line to virologic failure (VF can occur at any time from any time during the treatment phase from week 1 to week 14). Subjects who experience Virologic Failure will be followed up every 4 weeks until the viral load suppression is achieved (i.e., plasma HIV-1 RNA levels to return back to <50 copies/mL)
Time Frame: From baseline to virologic failure (VF occurring at any time from Week 1 to Week 12 or virologic failure which ever comes first)
Population: Per Protocol
Measure: Count of Participants; unit: Participants
Groups:
- PRO 140 350 mg: PRO 140 350 mg weekly SC injection
Arm/Group | PRO 140 350 mg
Number analyzed (Participants) | 41
Participants
  T1 (Week 1): Poor | 0
  T1 (Week 1): Fair | 1
  T1 (Week 1): Good | 6
  T1 (Week 1): Very Good | 10
  T1 (Week 1): Excellent | 13
  T1 (Week 1): Missing | 11
  T4 (Week 4): Poor | 0
  T4 (Week 4): Fair | 1
  T4 (Week 4): Good | 6
  T4 (Week 4): Very Good | 11
  T4 (Week 4): Excellent | 12
  T4 (Week 4): Missing | 11
  T8 (Week 8): Poor | 1
  T8 (Week 8): Fair | 2
  T8 (Week 8): Good | 6
  T8 (Week 8): Very Good | 9
  T8 (Week 8): Excellent | 9
  T8 (Week 8): Missing | 14
  T12 (Week 12): Poor | 0
  T12 (Week 12): Fair | 2
  T12 (Week 12): Good | 2
  T12 (Week 12): Very Good | 12
  T12 (Week 12): Excellent | 5
  T12 (Week 12): Missing | 20
  VF (Virologic Failure): Poor | 0
  VF (Virologic Failure): Fair | 0
  VF (Virologic Failure): Good | 3
  VF (Virologic Failure): Very Good | 3
  VF (Virologic Failure): Excellent | 1
  VF (Virologic Failure): Missing | 34

8. Secondary Outcome: Q2 QOL Current State of Health
Description: Subjects will rate their current state of health via Visual Analog Scale (VAS) using the line as a guide, with 0 as death or worst possible health and 100 as perfect or best possible health. A higher score indicates best outcome. Subjects may experience Virologic Failure (VF) any time during the treatment phase from week 1 to week 14. Subjects who experience VF will be followed up every 4 weeks until the viral load suppression is achieved (i.e., plasma HIV-1 RNA levels to return back to <50 copies/mL)
Time Frame: From week 1 through treatment weeks 4, 8, 12 or VF visit
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- PRO 140 350mg: PRO 140 350mg weekly SQ injection.: CCR5 Antagonist
Arm/Group | PRO 140 350mg
Number analyzed (Participants) | 30
score on a scale
  T1 (Week 1) | 82.3 (16.4)
  T4 (Week 4) | 83.8 (16.2)
  T8 (Week 8): number analyzed (Participants) | 27
  T8 (Week 8) | 80.9 (18.0)
  T12 (Week 12): number analyzed (Participants) | 21
  T12 (Week 12) | 84.9 (17.3)
  VF (Viral Failure): number analyzed (Participants) | 7
  VF (Viral Failure) | 78.0 (15.8)

9. Other Pre Specified Outcome: Injection Site Reaction - Pain (Site 1)
Description: Injection site reaction pain assessment @ injection site 1. Each subject received half the total dose of the IP into two separate injection sites. (injection site 1 and injection site 2) at each treatment visit. The information is reported under separate outcomes measures for each injection site.
Time Frame: From initiation of PRO 140 monotherapy through week 14
Population: Safety
Measure: Count of Participants; unit: Participants
Groups:
- PRO 140 350 mg Weekly SQ Injection: PRO 140 350mg weekly SQ injection.: CCR5 Antagonist
Arm/Group | PRO 140 350 mg Weekly SQ Injection
Number analyzed (Participants) | 43
Participants
  T1 (Week 1): absent | 43
  T1 (Week 1): present | 0
  T2 (Week 2): absent | 43
  T2 (Week 2): present | 0
  T3 (Week 3): absent | 43
  T3 (Week 3): present | 0
  T4 (Week 4): absent | 43
  T4 (Week 4): present | 0
  T5 (Week 5): absent | 43
  T5 (Week 5): present | 0
  T6 (Week 6): absent | 43
  T6 (Week 6): present | 0
  T7 (Week 7): number analyzed (Participants) | 41
  T7 (Week 7): absent | 41
  T7 (Week 7): present | 0
  T8 (Week 8): number analyzed (Participants) | 36
  T8 (Week 8): absent | 36
  T8 (Week 8): present | 0
  T9 (Week 9): number analyzed (Participants) | 33
  T9 (Week 9): absent | 33
  T9 (Week 9): present | 0
  T10 (Week 10): number analyzed (Participants) | 29
  T10 (Week 10): absent | 29
  T10 (Week 10): present | 0
  T11 (Week 11): number analyzed (Participants) | 29
  T11 (Week 11): absent | 29
  T11 (Week 11): present | 0
  T12 (Week 12): number analyzed (Participants) | 27
  T12 (Week 12): absent | 27
  T12 (Week 12): present | 0
  T13 (Week 13): number analyzed (Participants) | 23
  T13 (Week 13): absent | 22
  T13 (Week 13): present | 1
  T14 (Week 14): number analyzed (Participants) | 6
  T14 (Week 14): absent | 6
  T14 (Week 14): present | 0

10. Other Pre Specified Outcome: Injection Site Reaction - Pain (Site 2)
Description: Injection site reaction pain assessment @ injection site 2. Each subject received half the total dose of the IP into two separate injection sites. (injection site 1 and injection site 2) at each treatment visit. The information is reported under separate outcomes measures for each injection site.
Time Frame: From initiation of PRO 140 monotherapy through week 14
Population: safety population
Measure: Count of Participants; unit: Participants
Arm/Group | PRO 140 350mg
Number analyzed (Participants) | 43
Participants
  T1 (Week 1): absent | 43
  T1 (Week 1): present | 0
  T2 (Week 2): absent | 43
  T2 (Week 2): present | 0
  T3 ( Week 3): absent | 43
  T3 ( Week 3): present | 0
  T4 (Week 4): absent | 43
  T4 (Week 4): present | 0
  T5 (Week 5): absent | 43
  T5 (Week 5): present | 0
  T6 (Week 6): absent | 43
  T6 (Week 6): present | 0
  T7 (Week 7): number analyzed (Participants) | 41
  T7 (Week 7): absent | 41
  T7 (Week 7): present | 0
  T8 (Week 8): number analyzed (Participants) | 36
  T8 (Week 8): absent | 36
  T8 (Week 8): present | 0
  T9 (Week 9): number analyzed (Participants) | 29
  T9 (Week 9): absent | 29
  T9 (Week 9): present | 0
  T10 (Week 10): number analyzed (Participants) | 29
  T10 (Week 10): absent | 29
  T10 (Week 10): present | 0
  T11 (Week 11): number analyzed (Participants) | 29
  T11 (Week 11): absent | 29
  T11 (Week 11): present | 0
  T12 (Week 12): number analyzed (Participants) | 27
  T12 (Week 12): absent | 27
  T12 (Week 12): present | 0
  T13 (Week 13): number analyzed (Participants) | 23
  T13 (Week 13): absent | 23
  T13 (Week 13): present | 0
  T14 ( Week 14): number analyzed (Participants) | 6
  T14 ( Week 14): absent | 6
  T14 ( Week 14): present | 0

11. Other Pre Specified Outcome: Injection Site Reaction - Injection Site Status (Site 1)
Description: Summary of injection site reaction assessment - Injection site status @ injection site 1. Each subject received half the total dose of the IP into two separate injection sites. (injection site 1 and injection site 2) at each treatment visit. The information is reported under separate outcomes measures for each injection site.
Time Frame: From initiation of PRO 140 monotherapy through week 14
Population: safety
Measure: Count of Participants; unit: Participants
Arm/Group | PRO 140 350mg
Number analyzed (Participants) | 43
Participants
  T1 (Week 1): Normal | 43
  T1 (Week 1): abnormal | 0
  T2 (Week 2): Normal | 43
  T2 (Week 2): abnormal | 0
  T3 (Week 3): Normal | 43
  T3 (Week 3): abnormal | 0
  T4 (Week 4): Normal | 43
  T4 (Week 4): abnormal | 0
  T5 (Week 5): Normal | 43
  T5 (Week 5): abnormal | 0
  T6 (Week 6): Normal | 42
  T6 (Week 6): abnormal | 1
  T7 (Week 7): number analyzed (Participants) | 41
  T7 (Week 7): Normal | 41
  T7 (Week 7): abnormal | 0
  T8 (Week 8): number analyzed (Participants) | 36
  T8 (Week 8): Normal | 36
  T8 (Week 8): abnormal | 0
  T9 (Week 9): number analyzed (Participants) | 33
  T9 (Week 9): Normal | 33
  T9 (Week 9): abnormal | 0
  T10 (Week 10): number analyzed (Participants) | 29
  T10 (Week 10): Normal | 29
  T10 (Week 10): abnormal | 0
  T11 (Week 11): number analyzed (Participants) | 29
  T11 (Week 11): Normal | 29
  T11 (Week 11): abnormal | 0
  T12 (Week 12): number analyzed (Participants) | 27
  T12 (Week 12): Normal | 27
  T12 (Week 12): abnormal | 0
  T13 (Week 13): number analyzed (Participants) | 23
  T13 (Week 13): Normal | 23
  T13 (Week 13): abnormal | 0
  T14 (Week 14): number analyzed (Participants) | 6
  T14 (Week 14): Normal | 6
  T14 (Week 14): abnormal | 0

12. Other Pre Specified Outcome: Injection SIte Reaction - Injection Site Status (Site 2)
Description: Summary of injection site reaction assessment - Injection site status @ injection site 2. Each subject received half the total dose of the IP into two separate injection sites. (injection site 1 and injection site 2) at each treatment visit. The information is reported under separate outcomes measures for each injection site.
Time Frame: From initiation of PRO 140 monotherapy through week 14
Population: safety
Measure: Count of Participants; unit: Participants
Arm/Group | PRO 140 350 mg Weekly SQ Injection
Number analyzed (Participants) | 43
Participants
  T1 (Week 1): Normal | 43
  T1 (Week 1): Abnormal | 0
  T2 (Week 2): Normal | 43
  T2 (Week 2): Abnormal | 0
  T3 (Week 3): Normal | 43
  T3 (Week 3): Abnormal | 0
  T4 (Week 4): Normal | 43
  T4 (Week 4): Abnormal | 0
  T5 (Week 5): Normal | 43
  T5 (Week 5): Abnormal | 0
  T6 (Week 6): Normal | 42
  T6 (Week 6): Abnormal | 1
  T7 (Week 7): number analyzed (Participants) | 41
  T7 (Week 7): Normal | 41
  T7 (Week 7): Abnormal | 0
  T8 (Week 8): number analyzed (Participants) | 36
  T8 (Week 8): Normal | 36
  T8 (Week 8): Abnormal | 0
  T9 (Week 9): number analyzed (Participants) | 33
  T9 (Week 9): Normal | 33
  T9 (Week 9): Abnormal | 0
  T10 (Week 10): number analyzed (Participants) | 29
  T10 (Week 10): Normal | 29
  T10 (Week 10): Abnormal | 0
  T11 (Week 11): number analyzed (Participants) | 29
  T11 (Week 11): Normal | 29
  T11 (Week 11): Abnormal | 0
  T12 (Week 12): number analyzed (Participants) | 27
  T12 (Week 12): Normal | 27
  T12 (Week 12): Abnormal | 0
  T13 (Week 13): number analyzed (Participants) | 23
  T13 (Week 13): Normal | 23
  T13 (Week 13): Abnormal | 0
  T14 (Week 14): number analyzed (Participants) | 6
  T14 (Week 14): Normal | 6
  T14 (Week 14): Abnormal | 0

13. Other Pre Specified Outcome: Injection Site Reaction - Pruritus With Injection (Site 1)
Description: Summary of injection site reaction assessment - Pruritus with injection @Site 1. Each subject received half the total dose of the IP into two separate injection sites. (injection site 1 and injection site 2) at each treatment visit. The information is reported under separate outcomes measures for each injection site.
Time Frame: From initiation of PRO 140 monotherapy through week 14
Population: safety
Measure: Count of Participants; unit: Participants
Arm/Group | PRO 140 350mg
Number analyzed (Participants) | 43
Participants
  T1 (Week 1): Absent | 43
  T1 (Week 1): Present | 0
  T2 (Week 2): Absent | 42
  T2 (Week 2): Present | 1
  T3 (Week 3): Absent | 43
  T3 (Week 3): Present | 0
  T4 (Week 4): Absent | 43
  T4 (Week 4): Present | 0
  T5 (Week 5): Absent | 43
  T5 (Week 5): Present | 0
  T6 (Week 6): Absent | 43
  T6 (Week 6): Present | 0
  T7 (Week 7): number analyzed (Participants) | 41
  T7 (Week 7): Absent | 41
  T7 (Week 7): Present | 0
  T8 (Week 8): number analyzed (Participants) | 36
  T8 (Week 8): Absent | 36
  T8 (Week 8): Present | 0
  T9 (Week 9): number analyzed (Participants) | 33
  T9 (Week 9): Absent | 33
  T9 (Week 9): Present | 0
  T10 (Week 10): number analyzed (Participants) | 29
  T10 (Week 10): Absent | 29
  T10 (Week 10): Present | 0
  T11 (Week 11): number analyzed (Participants) | 29
  T11 (Week 11): Absent | 29
  T11 (Week 11): Present | 0
  T12 (Week 12): number analyzed (Participants) | 27
  T12 (Week 12): Absent | 27
  T12 (Week 12): Present | 0
  T13 (Week 13): number analyzed (Participants) | 23
  T13 (Week 13): Absent | 23
  T13 (Week 13): Present | 0
  T14 (Week 14): number analyzed (Participants) | 6
  T14 (Week 14): Absent | 6
  T14 (Week 14): Present | 0

14. Other Pre Specified Outcome: Injection Site Reaction - Pruritus With Injection (Site 2)
Description: Summary of injection site reaction assessment - Pruritus with injection @ Site 2. Each subject received half the total dose of the IP into two separate injection sites. (injection site 1 and injection site 2) at each treatment visit. The information is reported under separate outcomes measures for each injection site.
Time Frame: From initiation of PRO 140 monotherapy through week14
Population: safety
Measure: Count of Participants; unit: Participants
Arm/Group | PRO 140 350mg
Number analyzed (Participants) | 43
Participants
  T1 (Week 1): Absent | 43
  T1 (Week 1): Present | 0
  T2 (Week 2): Absent | 42
  T2 (Week 2): Present | 1
  T3 (Week 3): Absent | 43
  T3 (Week 3): Present | 0
  T4 (Week 4): Absent | 43
  T4 (Week 4): Present | 0
  T5 (Week 5): Absent | 43
  T5 (Week 5): Present | 0
  T6 (Week 6): Absent | 43
  T6 (Week 6): Present | 0
  T7 (Week 7): Absent | 41
  T7 (Week 7): Present | 2
  T8 (Week 8): number analyzed (Participants) | 36
  T8 (Week 8): Absent | 36
  T8 (Week 8): Present | 0
  T9 (Week 9): number analyzed (Participants) | 33
  T9 (Week 9): Absent | 33
  T9 (Week 9): Present | 0
  T10 (Week 10): number analyzed (Participants) | 29
  T10 (Week 10): Absent | 29
  T10 (Week 10): Present | 0
  T11 (Week 11): number analyzed (Participants) | 29
  T11 (Week 11): Absent | 29
  T11 (Week 11): Present | 0
  T12 (Week 12): number analyzed (Participants) | 27
  T12 (Week 12): Absent | 27
  T12 (Week 12): Present | 0
  T13 (Week 13): number analyzed (Participants) | 23
  T13 (Week 13): Absent | 23
  T13 (Week 13): Present | 0
  T14 (Week 14): number analyzed (Participants) | 6
  T14 (Week 14): Absent | 6
  T14 (Week 14): Present | 0

15. Other Pre Specified Outcome: Injection Site Reaction - Bleeding Site 1
Description: Summary of injection site reaction assessment - bleeding @ Site 1. Each subject received half the total dose of the IP into two separate injection sites. (injection site 1 and injection site 2) at each treatment visit. The information is reported under separate outcomes measures for each injection site.
Time Frame: From initiation of PRO 140 monotherapy through week 14
Population: safety
Measure: Count of Participants; unit: Participants
Arm/Group | PRO 140 350mg
Number analyzed (Participants) | 43
Participants
  T1 (Week 1): Absent | 43
  T1 (Week 1): Present | 0
  T2 (Week 2): Absent | 43
  T2 (Week 2): Present | 0
  T3 (Week 3): Absent | 43
  T3 (Week 3): Present | 0
  T4 (Week 4): Absent | 43
  T4 (Week 4): Present | 0
  T5 (Week 5): Absent | 43
  T5 (Week 5): Present | 0
  T6 (Week 6): Absent | 43
  T6 (Week 6): Present | 0
  T7 (Week 7): number analyzed (Participants) | 41
  T7 (Week 7): Absent | 41
  T7 (Week 7): Present | 0
  T8 (Week 8): number analyzed (Participants) | 36
  T8 (Week 8): Absent | 36
  T8 (Week 8): Present | 0
  T9 (Week 9): number analyzed (Participants) | 33
  T9 (Week 9): Absent | 33
  T9 (Week 9): Present | 0
  T10 (Week 10): number analyzed (Participants) | 29
  T10 (Week 10): Absent | 29
  T10 (Week 10): Present | 0
  T11 (Week 11): number analyzed (Participants) | 29
  T11 (Week 11): Absent | 29
  T11 (Week 11): Present | 0
  T12 (Week 12): number analyzed (Participants) | 27
  T12 (Week 12): Absent | 27
  T12 (Week 12): Present | 0
  T13 (Week 13): number analyzed (Participants) | 23
  T13 (Week 13): Absent | 23
  T13 (Week 13): Present | 0
  T14 (Week 14): number analyzed (Participants) | 6
  T14 (Week 14): Absent | 6
  T14 (Week 14): Present | 0

16. Other Pre Specified Outcome: Injection Site Reaction - Bleeding - Site 2
Description: Summary of injection site reaction assessment - bleeding @ Site 2. Each subject received half the total dose of the IP into two separate injection sites. (injection site 1 and injection site 2) at each treatment visit. The information is reported under separate outcomes measures for each injection site.
Time Frame: From initiation of PRO 140 monotherapy through week14
Population: safety
Measure: Count of Participants; unit: Participants
Arm/Group | PRO 140 350mg
Number analyzed (Participants) | 43
Participants
  T1 (Week 1): Absent | 43
  T1 (Week 1): Present | 0
  T2 (Week 2): Absent | 43
  T2 (Week 2): Present | 0
  T3 (Week 3): Absent | 43
  T3 (Week 3): Present | 0
  T4 (Week 4): Absent | 43
  T4 (Week 4): Present | 0
  T5 (Week 5): number analyzed (Participants) | 42
  T5 (Week 5): Absent | 42
  T5 (Week 5): Present | 0
  T6 (Week 6): number analyzed (Participants) | 42
  T6 (Week 6): Absent | 42
  T6 (Week 6): Present | 0
  T7 (Week 7): number analyzed (Participants) | 41
  T7 (Week 7): Absent | 41
  T7 (Week 7): Present | 0
  T8 (Week 8): number analyzed (Participants) | 36
  T8 (Week 8): Absent | 36
  T8 (Week 8): Present | 0
  T9 (Week 9): number analyzed (Participants) | 33
  T9 (Week 9): Absent | 33
  T9 (Week 9): Present | 0
  T10 (Week 10): number analyzed (Participants) | 29
  T10 (Week 10): Absent | 29
  T10 (Week 10): Present | 0
  T11 (Week 11): number analyzed (Participants) | 29
  T11 (Week 11): Absent | 29
  T11 (Week 11): Present | 0
  T12 (Week 12): number analyzed (Participants) | 27
  T12 (Week 12): Absent | 26
  T12 (Week 12): Present | 1
  T13 (Week 13): number analyzed (Participants) | 23
  T13 (Week 13): Absent | 23
  T13 (Week 13): Present | 0
  T14 (Week 14): number analyzed (Participants) | 6
  T14 (Week 14): Absent | 6
  T14 (Week 14): Present | 0

17. Other Pre Specified Outcome: Injection Site Reaction - Drug Absorption - Site 1
Description: Summary of injection site reaction assessment - drug absorption @ Site 1. Each subject received half the total dose of the IP into two separate injection sites. (injection site 1 and injection site 2) at each treatment visit. The information is reported under separate outcomes measures for each injection site.
Time Frame: From initiation of PRO 140 monotherapy through week14
Population: safety
Measure: Count of Participants; unit: Participants
Arm/Group | PRO 140 350mg
Number analyzed (Participants) | 43
Participants
  T1 (Week 1): Normal | 43
  T1 (Week 1): Abnormal | 0
  T2 (Week 2): Normal | 43
  T2 (Week 2): Abnormal | 0
  T3 (Week 3): Normal | 43
  T3 (Week 3): Abnormal | 0
  T4 (Week 4): Normal | 43
  T4 (Week 4): Abnormal | 0
  T5 (Week 5): Normal | 43
  T5 (Week 5): Abnormal | 0
  T6 (Week 6): Normal | 43
  T6 (Week 6): Abnormal | 0
  T7 (Week 7): number analyzed (Participants) | 41
  T7 (Week 7): Normal | 41
  T7 (Week 7): Abnormal | 0
  T8 (Week 8): number analyzed (Participants) | 36
  T8 (Week 8): Normal | 36
  T8 (Week 8): Abnormal | 0
  T9 (Week 9): number analyzed (Participants) | 33
  T9 (Week 9): Normal | 33
  T9 (Week 9): Abnormal | 0
  T10 (Week 10): number analyzed (Participants) | 29
  T10 (Week 10): Normal | 29
  T10 (Week 10): Abnormal | 0
  T11 (Week 11): number analyzed (Participants) | 29
  T11 (Week 11): Normal | 29
  T11 (Week 11): Abnormal | 0
  T12 (Week 12): number analyzed (Participants) | 27
  T12 (Week 12): Normal | 27
  T12 (Week 12): Abnormal | 0
  T13 (Week 13): number analyzed (Participants) | 23
  T13 (Week 13): Normal | 23
  T13 (Week 13): Abnormal | 0
  T14 (Week 14): number analyzed (Participants) | 6
  T14 (Week 14): Normal | 6
  T14 (Week 14): Abnormal | 0

18. Other Pre Specified Outcome: Injection Site Reaction - Drug Absorption - Site 2
Description: Summary of injection site reaction assessment - drug absorption @ Site 2. Each subject received half the total dose of the IP into two separate injection sites. (injection site 1 and injection site 2) at each treatment visit. The information is reported under separate outcomes measures for each injection site.
Time Frame: From initiation of PRO 140 monotherapy through week 14
Population: safety
Measure: Count of Participants; unit: Participants
Arm/Group | PRO 140 350mg
Number analyzed (Participants) | 43
Participants
  T1 (Week 1): Normal | 43
  T1 (Week 1): Abnormal | 0
  T2 (Week 2): Normal | 43
  T2 (Week 2): Abnormal | 0
  T3 (Week 3): Normal | 43
  T3 (Week 3): Abnormal | 0
  T4 (Week 4): Normal | 43
  T4 (Week 4): Abnormal | 0
  T5 (Week 5): Normal | 43
  T5 (Week 5): Abnormal | 0
  T6 (Week 6): Normal | 43
  T6 (Week 6): Abnormal | 0
  T7 (Week 7): number analyzed (Participants) | 41
  T7 (Week 7): Normal | 41
  T7 (Week 7): Abnormal | 0
  T8 (Week 8): number analyzed (Participants) | 36
  T8 (Week 8): Normal | 36
  T8 (Week 8): Abnormal | 0
  T9 (Week 9): number analyzed (Participants) | 33
  T9 (Week 9): Normal | 33
  T9 (Week 9): Abnormal | 0
  T10 (Week 10): number analyzed (Participants) | 29
  T10 (Week 10): Normal | 29
  T10 (Week 10): Abnormal | 0
  T11 (Week 11): number analyzed (Participants) | 29
  T11 (Week 11): Normal | 29
  T11 (Week 11): Abnormal | 0
  T12 (Week 12): number analyzed (Participants) | 27
  T12 (Week 12): Normal | 27
  T12 (Week 12): Abnormal | 0
  T13 (Week 13): number analyzed (Participants) | 23
  T13 (Week 13): Normal | 23
  T13 (Week 13): Abnormal | 0
  T14 (Week 14): number analyzed (Participants) | 6
  T14 (Week 14): Normal | 6
  T14 (Week 14): Abnormal | 0

19. Other Pre Specified Outcome: Injection Site Reaction - Pain Post Injection - Site 1
Description: Summary of injection site pain assessment (VAS) post injection mean change from baseline. Subject-perceived injection site pain was assessed using the Pain Visual Analog Scale (VAS) post study treatment administration assessing average pain. Higher score is worse outcome. Each subject received half the total dose of the IP into two separate injection sites. (injection site 1 and injection site 2) at each treatment visit. The information is reported under separate outcomes measures for each injection site.
Time Frame: From initiation of PRO 140 monotherapy through week 14
Population: Safety
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PRO 140 350mg
Number analyzed (Participants) | 43
score on a scale
  T1 (Week 1): number analyzed (Participants) | 12
  T1 (Week 1) | 18.4 (16.1)
  T2 (Week 2): number analyzed (Participants) | 12
  T2 (Week 2) | -3.9 (8.6)
  T3 (Week 3): number analyzed (Participants) | 11
  T3 (Week 3) | -7.9 (11.4)
  T4 (Week 4): number analyzed (Participants) | 12
  T4 (Week 4) | -2.5 (14.2)
  T5 (Week 5): number analyzed (Participants) | 12
  T5 (Week 5) | -12.8 (13.9)
  T6 (Week 6): number analyzed (Participants) | 12
  T6 (Week 6) | -6.8 (16.7)
  T7 (Week 7): number analyzed (Participants) | 11
  T7 (Week 7) | -13.5 (13.9)
  T8 (Week 8): number analyzed (Participants) | 8
  T8 (Week 8) | -16.6 (14.8)
  T9 (Week 9): number analyzed (Participants) | 8
  T9 (Week 9) | -15.0 (14.2)
  T10 (Week 10): number analyzed (Participants) | 6
  T10 (Week 10) | -17.2 (12.3)
  T11 (Week 11): number analyzed (Participants) | 6
  T11 (Week 11) | -24.0 (18.1)
  T12 (Week 12): number analyzed (Participants) | 6
  T12 (Week 12) | -22.0 (18.4)
  T13 (Week 13): number analyzed (Participants) | 5
  T13 (Week 13) | -17.0 (15.6)
  T14 (Week 14): number analyzed (Participants) | 5
  T14 (Week 14) | -22.0 (19.1)

20. Other Pre Specified Outcome: Injection Site Reaction - Pain Post Injection - Site 2
Description: Summary of injection site pain assessment (VAS) post injection @ Site 2. Subject-perceived injection site pain was assessed using the Pain Visual Analog Scale (VAS) post study treatment administration assessing average pain. A higher score is a worse outcome. Each subject received half the total dose of the IP into two separate injection sites. (injection site 1 and injection site 2) at each treatment visit. The information is reported under separate outcomes measures for each injection site.
Time Frame: From initiation of PRO 140 monotherapy through week 14
Population: Safety
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PRO 140 350mg
Number analyzed (Participants) | 43
score on a scale
  T1 (Week 1): number analyzed (Participants) | 12
  T1 (Week 1) | 17.4 (15.2)
  T2 (Week 2): number analyzed (Participants) | 12
  T2 (Week 2) | -2.0 (14.2)
  T3 (Week 3): number analyzed (Participants) | 12
  T3 (Week 3) | -4.8 (11.8)
  T4 (Week 4): number analyzed (Participants) | 12
  T4 (Week 4) | -7.8 (12.2)
  T5 (Week 5): number analyzed (Participants) | 12
  T5 (Week 5) | -8.8 (15.7)
  T6 (Week 6): number analyzed (Participants) | 12
  T6 (Week 6) | -7.2 (17.6)
  T7 (Week 7): number analyzed (Participants) | 11
  T7 (Week 7) | -10.4 (14.8)
  T8 (Week 8): number analyzed (Participants) | 8
  T8 (Week 8) | -13.0 (15.9)
  T9 (Week 9): number analyzed (Participants) | 8
  T9 (Week 9) | -14.6 (16.0)
  T10 (Week 10): number analyzed (Participants) | 6
  T10 (Week 10) | -10.7 (9.1)
  T11 (Week 11): number analyzed (Participants) | 6
  T11 (Week 11) | -14.7 (13.3)
  T12 (Week 12): number analyzed (Participants) | 6
  T12 (Week 12) | -15.2 (14.8)
  T13 (Week 13): number analyzed (Participants) | 5
  T13 (Week 13) | -10.0 (10.3)
  T14 (Week 14): number analyzed (Participants) | 5
  T14 (Week 14) | -13.8 (18.5)

21. Other Pre Specified Outcome: Injection Site Reaction - Pain Pre Injection - Site 1
Description: Summary of injection site pain assessment (VAS) pre injection @ Site 1 Subject-perceived injection site pain was assessed using the Pain Visual Analog Scale (VAS) prior to study treatment administration assessing average pain since last treatment. Higher score is a worse outcome. Each subject received half the total dose of the IP into two separate injection sites. (injection site 1 and injection site 2) at each treatment visit. The information is reported under separate outcomes measures for each injection site.
Time Frame: From week 2 through week 14
Population: Safety
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PRO 140 350mg
Number analyzed (Participants) | 43
score on a scale
  T2 (Week 2): number analyzed (Participants) | 30
  T2 (Week 2) | 0.0 (0.0)
  T3 (Week 3): number analyzed (Participants) | 30
  T3 (Week 3) | 2.8 (8.4)
  T4 (Week 4): number analyzed (Participants) | 30
  T4 (Week 4) | 1.7 (6.6)
  T5 (Week 5): number analyzed (Participants) | 30
  T5 (Week 5) | 2.2 (4.2)
  T6 (Week 6): number analyzed (Participants) | 30
  T6 (Week 6) | 1.6 (4.2)
  T7 (Week 7): number analyzed (Participants) | 29
  T7 (Week 7) | 1.0 (4.0)
  T8 (Week 8): number analyzed (Participants) | 27
  T8 (Week 8) | 0.9 (3.6)
  T9 (Week 9): number analyzed (Participants) | 24
  T9 (Week 9) | 1.6 (4.1)
  T10 (Week 10): number analyzed (Participants) | 22
  T10 (Week 10) | 1.5 (5.9)
  T11 (Week 11): number analyzed (Participants) | 22
  T11 (Week 11) | 1.3 (4.7)
  T12 (Week 12): number analyzed (Participants) | 20
  T12 (Week 12) | 0.5 (4.1)
  T13 (Week 13): number analyzed (Participants) | 16
  T13 (Week 13) | 0.6 (1.3)
  T14 (Week 14): number analyzed (Participants) | 1
  T14 (Week 14) | 0.0 (NA) — The SD is not computed because n=1

22. Other Pre Specified Outcome: Injection Site Reaction - Pain Pre Injection - Site 2
Description: Summary of injection site pain assessment (VAS) pre injection @ Site 2. Subject-perceived injection site pain was assessed using the Pain Visual Analog Scale (VAS) prior to study treatment administration assessing average pain since last treatment. Higher score is a worse outcome. Each subject received half the total dose of the IP into two separate injection sites. (injection site 1 and injection site 2) at each treatment visit. The information is reported under separate outcomes measures for each injection site.
Time Frame: From week 2 through week 14
Population: Safety
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PRO 140 350mg
Number analyzed (Participants) | 43
score on a scale
  T2 (Week 2): number analyzed (Participants) | 30
  T2 (Week 2) | 0.0 (0.0)
  T3 (Week 3): number analyzed (Participants) | 30
  T3 (Week 3) | 2.4 (9.2)
  T4 (Week 4): number analyzed (Participants) | 30
  T4 (Week 4) | 4.8 (19.9)
  T5 (Week 5): number analyzed (Participants) | 30
  T5 (Week 5) | 2.1 (7.1)
  T6 (Week 6): number analyzed (Participants) | 30
  T6 (Week 6) | 2.0 (7.1)
  T7 (Week 7): number analyzed (Participants) | 29
  T7 (Week 7) | 0.8 (6.9)
  T8 (Week 8): number analyzed (Participants) | 27
  T8 (Week 8) | 1.1 (6.5)
  T9 (Week 9): number analyzed (Participants) | 24
  T9 (Week 9) | 1.9 (7.2)
  T10 (Week 10): number analyzed (Participants) | 22
  T10 (Week 10) | 1.7 (8.5)
  T11 (Week 11): number analyzed (Participants) | 22
  T11 (Week 11) | 1.4 (7.7)
  T12 (Week 12): number analyzed (Participants) | 20
  T12 (Week 12) | 0.1 (5.3)
  T13 (Week 13): number analyzed (Participants) | 16
  T13 (Week 13) | 0.4 (0.8)
  T14 (Week 14): number analyzed (Participants) | 1
  T14 (Week 14) | 0.0 (NA) — The SD was not computed because n=1

23. Other Pre Specified Outcome: Pro 140 Concentration
Description: Summary of Pro 140 Concentration. Subjects may experience Virologic Failure (VF) any time during the treatment phase from week 1 to week 14. Subjects who experience VF will be followed up every 4 weeks until the viral load suppression is achieved (i.e., plasma HIV-1 RNA levels to return back to <50 copies/mL).
Time Frame: At week 4, week 8, week 12 and viral failure visits
Population: Safety
Measure: Mean (Inter-Quartile Range); unit: ng/ml
Arm/Group | PRO 140 350mg
Number analyzed (Participants) | 43
ng/ml
  T4 (Week 4): number analyzed (Participants) | 26
  T4 (Week 4) | 18084 [8152 to 37318]
  T8 (Week 8): number analyzed (Participants) | 28
  T8 (Week 8) | 22010 [6965 to 41624]
  T12 (Week 12): number analyzed (Participants) | 21
  T12 (Week 12) | 26388 [11632 to 74414]
  VF (Viral Failure): number analyzed (Participants) | 9
  VF (Viral Failure) | 16258 [8133 to 26396]

ADVERSE EVENTS:
Time Frame: Adverse events were collected for a total of 18 weeks, from treatment visit 1 (Post Rx) to treatment visit T14 (Week 14) and through the follow up period, every 2 week for total of 4 weeks. The duration of follow-up depends on the status of viral load suppression. Subjects who experience Virologic Failure will be discontinued from the treatment phase and be followed up every 4 weeks until the viral load suppression is achieved (i.e., plasma HIV-1 RNA levels to return back to <50 copies/mL).
Groups:
- Leronlimab: Leronlimab Pro 140
Arm/Group | Leronlimab
All-Cause Mortality (participants affected / at risk) | 0/43
Serious Adverse Events (participants affected / at risk) | 1/43
Other Adverse Events (participants affected / at risk) | 7/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Leronlimab (N=43)
transient ischemic attack (Nervous system disorders) | 1 (1) — TIA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Leronlimab (N=43)
nasopharyngitis (Infections and infestations) | 4
Constipation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 4
nausea (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 4
Injection site pruritus (General disorders) | 4
Dizziness (Nervous system disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No